CLINICAL TRIAL: NCT06483802
Title: A Multicenter, Open-Label, Dose Escalation, Phase 1b Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of ASP2016 for Friedreich Ataxia Cardiomyopathy
Brief Title: A Study of ASP2016 in Adults Who Have Heart Disease Associated With Friedreich Ataxia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate decision to withdraw the trial at this time.
Sponsor: Astellas Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-CL-0101
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Friedreich Ataxia; Cardiomyopathy
Keywords: ASP2016; Friedreich Ataxia Cardiomyopathy; Frataxin; Friedreichs Ataxia; Heart; Gene Therapy
MeSH Terms: conditions — Friedreich Ataxia; Cardiomyopathies | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASP2016 (Experimental): Participants will receive a single dose of ASP2016. Participants will also receive daily prednisolone beginning 1 day prior to ASP2016 dose and for at least 16 weeks after ASP2016 dose, in order to suppress the immune response to ASP2016.
  Interventions: Genetic: ASP2016; Drug: Prednisolone

INTERVENTIONS:
Genetic: ASP2016 — Intravenous (IV) infusion
Drug: Prednisolone — Oral

SUMMARY:
Friedreich Ataxia is a rare condition that causes damage to the nervous system and muscles. People with Friedreich Ataxia have difficulty walking, lose sensation in their arms and legs, and have slurred speech. It can also affect the heart and many people with Friedrich Ataxia develop serious heart problems. Friedreich Ataxia is a genetic condition which means a faulty gene is passed down through families. This type of gene therapy treats a genetic condition by providing a healthy copy of the gene.

At the time this study started, there was no approved treatment for heart problems in people with Friedreich Ataxia.

In this study, ASP2016 is being tested in humans for the first time. The people taking part are adults with Friedreich Ataxia who have heart problems.

The main aims of the study are to check the safety of ASP2016 and how people cope with (tolerate) ASP2016. ASP2016 is given as a slow injection into a vein. This is called an infusion. People will also take tablets of a medicine called prednisolone. This is taken to stop the immune system interfering with ASP2016.

Each person in the study will be given 1 single infusion of ASP2016. Different small groups will receive lower or higher doses of ASP2016. Each person will stay overnight in the clinic for at least 1 night after their infusion.

For the first few months, people will visit the clinic regularly. There may be the option of home visits by a study nurse at some visits. At the 6-month and 12-month visits extra tests, procedures, and scans will be done. One of these is an ECHO (echocardiogram) scan. This is like an ultrasound scan for the heart. Another is an endomyocardial biopsy. A tiny piece of their heart tissue is removed (biopsy). A flexible hollow tube (catheter) goes into the blood vessels up to the heart. Then, a small device on the end of the catheter takes a tiny piece of heart tissue (about the size of a pencil tip). Another is a cardiac MRI. This takes pictures of the inside of the heart using a powerful magnet. Another is a cardiopulmonary exercise test (CPET). This involves moving a specially designed set of bicycle pedals using hands and arms. This will check how the lungs, heart and muscles are affected during exercise.

After the 12-month visit, people will visit the clinic every few months for up to a few years.

ELIGIBILITY:
Inclusion Criteria:

* Participant has both a clinical diagnosis of Friedreich ataxia (FA) and a documented history of genetic diagnosis of FA with either a guanine-adenine-adenine (GAA) trinucleotide repeat (TNR) expansion in intron 1 of both gene for frataxin (FXN) alleles or a GAA TNR expansion of intron 1 of one FXN allele and a pathogenic variant in the other FXN allele.
* Participant has a resting LVEF ≥ 40% and < 55% as measured at screening by ECHO.
* Participant has a body mass index range of 17.0 to 30.0 kg/m2.
* Participant agrees not to begin omaveloxolone treatment during the 52-week period after receiving study intervention.
* Participants on omaveloxolone, who opt to discontinue omaveloxolone, may enroll if they stop omaveloxolone for 3 weeks and pass study screening, including LFTs.
* Participants on omaveloxolone, who opt to stay on omaveloxolone will need to have been on it for a minimum of 3 months, with LFTs that pass diagnostic assessments exclusion criteria at screening and prior to dosing with ASP2016. Prior elevation(s) in AST/ALT associated with omaveloxolone use must be discussed with the sponsor medical monitor. If there is a liver function test (LFT) elevation after treatment, participant agrees to stop omaveloxolone treatment until 52 weeks.
* Participants on omaveloxolone will need to discontinue strong or moderate cytochrome P450 3A4 (CYP3A4) inducers and inhibitors.
* Woman of Child Bearing Potential (WOCBP) on omaveloxolone must use a nonhormonal, highly effective methods of contraception (e.g., nonhormonal intrauterine device system), as omaveloxolone may interfere with hormonal methods of contraception.

Exclusion Criteria:

* Participant has late-onset FA, defined as symptom onset after the age of 25 years.
* Participant is unable to complete cardiopulmonary exercise testing (CPET) procedure.
* Participant has a contraindication to endomyocardial biopsy or cardiac catheterization.
* Participant has a contraindication to cardiac magnetic resonance imaging (CMRI) with contrast, including hypersensitivity to gadolinium contrast agent, cardiac pacemaker or implantable cardiac defibrillator.
* Participant has an elevated titer of anti-AAV8 total antibodies, as determined by central testing.
* Participant has significant fibrosis on CMRI, defined as late gadolinium enhancement of > 15% left ventricular myocardial mass.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to month 60
  A TEAE is defined as an AE observed after starting administration of the study intervention.
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  Note: an AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Number of Participants with Serious Adverse Events (SAEs) | Up to month 60
  An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and other medically important events.
Number of participants with laboratory value abnormalities and/or AEs | Up to month 60
  Number of participants with potentially clinically significant laboratory values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to month 60
  Number of participants with potentially clinically significant ECG values.
Number of participants with physical exam value abnormalities and/or AEs | Up to month 60
  Number of participants with potentially clinically significant physical exam values.

SECONDARY OUTCOMES:
Change from baseline of frataxin protein level in cardiac tissue | Baseline, week 24 and week 52
  Frataxin protein level in cardiac tissue will be recorded from endomyocardial biopsies collected by cardiac catheterization.
Change from baseline of peak rate of oxygen consumption (VO2peak) | Baseline, week 24 and week 52
  VO2peak will be measured by upper extremity cardiopulmonary exercise testing (CPET).
Change from baseline of ventilatory anaerobic threshold (AT) | Baseline, week 24 and week 52
  AT will be measured by upper extremity CPET.
Change from baseline of ventilation (VE)/volume of exhaled carbon dioxide (VCO2) slope | Baseline, week 24 and week 52
  VE/VCO2 slope will be measured by upper extremity CPET.
Change from baseline of left ventricular ejection fraction (LVEF) | Baseline, week 24 and week 52
  LVEF will be measured by echocardiogram (ECHO).
Change from baseline of left ventricular mass index (LVMI) | Baseline, week 24 and week 52
  LVMI will be measured by ECHO.
Change from baseline of longitudinal cardiac strain | Baseline, week 24 and week 52
  Longitudinal cardiac strain will be measured by ECHO.
Change from baseline of vector copy number (VCN) | Baseline, week 24 and week 52
  VCN will be recorded from endomyocardial biopsies collected by cardiac catheterization.
Change from baseline of total antibody (TAb) to adeno-associated virus 8 (AAV8) | Baseline and up to week 52
  TAb to AAV8 will be recorded from serum samples collected.
Change from baseline of neutralizing antibody (NAb) to AAV8 | Baseline and up to week 52
  NAb to AAV8 will be recorded from serum samples collected.
Change from baseline of TAb to frataxin | Baseline and up to week 52
  TAb to frataxin will be recorded from serum samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Lead, Study Director — Astellas Pharma Global Development, Inc.

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.